CLINICAL TRIAL: NCT00610909
Title: Single-Site, Double-Blind, Flexible-Dose, Placebo-Controlled Study of the Efficacy, Tolerability, & Safety of Paroxetine - Controlled Release in the Treatment of Irritable Bowel Syndrome (IBS)
Brief Title: Paroxetine - Controlled Release in the Treatment of Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Greg Clary, M.D, Duke University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3611; IRB#3611
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2008-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Those in the active treatment group will receive doses of Paxil CR in increments of 12.5 mg daily for the first week and increased at 12.5 mg increments at visit weeks to a maximum of 50 mg daily, as determined by the investigator. The investigator will adjust dosage based on clinical response. Following the completion of the double-blind phase, patients on placebo and non-responders to the study drug will be tapered off the study drug back to 0 over 2 weeks, and they will be referred to their Primary Care Physician, Internist or Gastroenterologist to be prescribed treatment for Irritable Bowel Syndrome.
  Interventions: Drug: Paroxetine CR
- 2 (Placebo Comparator): Same shape placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine CR — Those in the active treatment group will receive doses of Paxil CR in increments of 12.5 mg daily for the first week and increased at 12.5 mg increments at visit weeks to a maximum of 50 mg daily, as determined by the investigator. The investigator will adjust dosage based on clinical response. Following the completion of the double-blind phase, patients on placebo and non-responders to the study drug will be tapered off the study drug back to 0 over 2 weeks, and they will be referred to their Primary Care Physician, Internist or Gastroenterologist to be prescribed treatment for Irritable Bowel Syndrome.
  Other Names: Paxil
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Irritable bowel syndrome (IBS) is an extremely common disorder in the U.S population, affecting somewhere between 9-22% based on community based studies. IBS has a chronic relapsing course and overlaps with other functional gastrointestinal disorders. It accounts for high direct medical expenses and indirect costs including a significant degree of absenteeism. Most studies have suggested that there is a slight predominance among women, especially those that have suffered some form of physical or sexual trauma. It has been estimated that up to 25-40% of patients seen by gastroenterologists' are affected by IBS, and that 70-90% of these patients may have a psychiatric comorbidity, most commonly major depression and panic disorder, but also including schizophrenia, double depression, dysthymia and alcohol abuse.

Abdominal pain and disturbance of bowel habits characterize the symptoms of IBS in the absence of demonstrable structural pathology. The diagnosis of IBS relies upon clinical criteria alone, as there is no "gold standard" in laboratory findings. The diagnosis is dependent upon identifying characteristic symptoms, and then differentiating IBS from other structural bowel disorders. Previously, the diagnosis of IBS was based upon a consortium recommendation that examined and defined diagnostic criteria for over 100 functional gastrointestinal disorders. These criteria became the most definitive in the area of functional disorders and are referred to as the Rome Criteria. During the time since this consensus, these criteria have been modified, and in 1999 became the foundation for the second set of diagnostic criteria by consensus, now referred to as the Rome II criteria. The revised Rome II criteria include only the first part of the original criteria, but now require the presence of two out of three symptoms relating abdominal pain to bowel symptoms.

We designed our study and a Randomized, double-blind, parallel-group, flexible-dose, placebo-controlled 12-week study.

DETAILED DESCRIPTION:
Primary and Secondary Efficacy Measures Primary

Change from baseline in:

• Mean composite pain scores (on IVRS) Secondary

Change from baseline in:

* Associated symptoms of IBS (diarrhea, constipation, incomplete emptying, etc.) scores
* IBS Quality of Life scores
* Clinical Global Impression scores of 1 or 2
* Beck Depression Inventory II
* Beck Anxiety Inventory

Safety Measures

Safety and tolerability will be assessed through:

* Recording of spontaneous adverse events throughout the screening, run-in, and treatment phases of the study
* Conducting the DOTES at defined points during the study

All subjects withdrawn from the study will be followed until complete resolution of adverse events.

Study Schedule This is a placebo-controlled, double-blinded prospective 12-week study examining the efficacy of paroxetine extended release form in patients with IBS. Patients meeting the Rome II criteria for IBS will be recruited from the Duke University Medical Center Division of Gastroenterology and from the community. Patients found to satisfy these criteria will be referred for enrollment into this study. The study will be explained and informed consent obtained. A detailed history about the gastrointestinal symptoms and a physical exam will be performed. Laboratory evaluations (CBC, chemistry, fecal occult blood, urinalysis and EKG) will be obtained.

All patients will undergo a MINI at baseline to diagnose any comorbid Axis I psychiatric disorders, and a physical and sexual abuse history will be elicited. The patients will then have 1 week of symptom charting using the Interactive Voice Response System (IVRS) to measure baseline severity of IBS symptoms. Following that, patients will receive a single-blind placebo for a 1 week period. Those patients having a >25% improvement in composite pain scores at the end of the placebo week or a CGI of 1 or 2 will be terminated from the study. Following the 1 week single-blind placebo lead-in, non-responders will be randomized to active drug or placebo for an additional period of 12 weeks. The patients will continue to fill out a daily symptom diary using the IVRS and, in addition, will have weekly visits (biweekly after week 4) to assess symptoms, side-effects, and improvement over the entire 12-week double-blind period. Those in the active treatment group will receive doses of Paxil CR in increments of 12.5 mg daily for the first week and increased at 12.5 mg increments at visit weeks to a maximum of 50 mg daily, as determined by the investigator. The investigator will adjust dosage based on clinical response. Following the completion of the double-blind phase, patients on placebo and non-responders to the study drug will be tapered off the study drug back to 0 over 2 weeks, and they will be referred to their Primary Care Physician, Internist or Gastroenterologist to be prescribed treatment for Irritable Bowel Syndrome. Patients on active drug (Paroxetine CR) who were successful responders during the double-blind phase will be eligible to continue on open label Paxil CR for an additional period of 6 months plus 2 weeks and will be followed on a monthly basis. They will complete the IVRS symptom diary for a week during each follow-up month for an additional 6 months. Those who completed the double-blind phase during the 1st half of the month (days 1-14) will complete the IVRS symptom diary for the first week beginning the 1st of the next month; those who completed the double-blind phase during the second half of the month (days 15-31) will complete the IVRS symptom diary for the first week beginning the 1st of the month following the next month. At the end of the 6-month period, study medication for these patients will be tapered back to 0 over 2 weeks, and they will be referred to their Primary Care Physician, Internist or Gastroenterologist to be prescribed treatment for the Irritable Bowel Syndrome. Placebo responders in the double-blind phase will not be eligible to enter the 6-month open label maintenance phase.

Clinical response will be measured in several ways. Abdominal pain severity will be measured with an ordinal scale rated from 1-9 (1=mild pain/discomfort, 9=very severe pain/discomfort). Abdominal pain frequency will be measured on a four-point scale (1=pain or discomfort present only occasionally, 2=pain or discomfort present less than half the day, 3= pain or discomfort present more than half the day, 4=pain or discomfort almost all day). The same ordinal scale will be used to quantify the distress or discomfort caused by feeling of incomplete evacuation, bloating or abdominal discomfort, and general level of stress or tension.

Sample Size Computation and Power Analysis Power considerations The calculations that follow are computed for the current design with an anticipated difference in pre-and post-treatment on the mean composite pain scores (on IVRS) of 25% (i.e. a reduction of score from 100 to 75). The means and standard deviations for this computation rely on our previous open-label studies of paroxetine and citalopram in IBS.

Assuming a strong effect size (0.5) of the primary variable (mean composite pain scores) and alpha set at 0.05, a projected sample size of 50 can detect the main effects with a power of greater than 0.95. If a lower effect size is assumed (0.4), a projected sample size of 55 can detect main effects with a power of approximately 0.94. Note that power may be reduced by attrition of the sample (i.e. dropouts) and also may be limited in testing secondary hypotheses where a further stratification of sample may be necessary (i.e. if the data is examined separately in men and women)

It may be more appropriate to have a sample size of 60 which allows for a 20% attrition rate and can still detect an effect size of 0.4 for the primary variable in the treatment-completer group with a power greater than 90.

Statistical analyses The study's main hypothesis is that paroxetine (Paxil CR) treatment will be more effective than placebo in reducing symptoms of IBS.

All statistical tests will be two sided at the 0.05 level of significance. Descriptive statistics will be used to provide a profile of demographic and outcome measures. Pearson product moment correlational analyses will be conducted to examine the relationships among variables. Baseline assessments between the two groups will be compared using chi square for categorical variables and independent t tests (two tailed) for continuous variables. Between group (medication/placebo) comparisons for primary and secondary variables will employ analysis of variance (ANOVA) with repeated measures. Assessments will be taken at baseline and end of week 1, 2, 3, 4, 6, 8, 10, and 12. Within group analyses (pre and end-of-treatment) will employ two tailed t tests.

To control for the possibility that current psychopathology might affect subject responding on interview and self-report instruments and otherwise modulate the treatment effects, the distribution of BDI-II and BAI scores and life time Axis I diagnoses in the placebo and control groups will be examined. The potential influence of any unequally distributed variables will be controlled via analyses-of covariance (ANCOVA) using the unequally distributed variables as covariates.

After the primary analysis other exploratory analyses will be conducted to test potential hypotheses for further studies.

ELIGIBILITY:
Inclusion Criteria

Each patient must satisfy all the following criteria before entry into the study:

1. Patients must have given their written informed consent to enter the study (after verification of the diagnosis criteria).
2. Male or female patients, aged 18 to 75 years of age at last birthday.

   Female patients of child-bearing potential must use one of the following methods of contraception for the duration of the study:
   * Oral contraceptive (combined or progesterone only)
   * Parenteral progesterone-only contraceptive (e.g. Norplant®, Depo-Provera®)
   * Intra-uterine device
   * Double barrier method of contraceptive (e.g. condom plus spermicide, condom plus diaphragm, etc.) Female patients of child-bearing potential will be defined as those who are not post-menopausal or those who have not undergone a hysterectomy or surgical sterilization. (Note: to be considered post-menopausal, a woman would have to be naturally free of menses for at least 2 years).
3. Patients presenting with Irritable Bowel Syndrome as defined by the modified Rome II Criteria:

   At least 12 weeks, which need not be consecutive, in the preceding 12 months of abdominal discomfort or pain that has two of three features:
   * Relieved with defecation; and/or
   * Onset associated with a change in frequency of stool; and/or
   * Onset associated with a change in form (appearance) of stool.

   The following symptoms cumulatively support the diagnosis of IBS:
   * Abnormal stool frequency
   * Abnormal stool form
   * Abnormal stool passage
   * Passage of mucus
   * Bloating or feeling of abdominal distention

   In order to proceed into the double-blind phase of the study, patients must have recorded at least 5 days' data for abdominal pain and Overall Assessment of symptoms on the IVRS during the placebo run-in period. In addition, the patient must demonstrate a <25% improvement in composite pain scores in placebo run-in period as compared to screening week.
4. Patients who have experienced symptoms of IBS for a duration of greater than one year (from the date of the Screening visit) and for whom this is documented in the medical notes.
5. Patients must be willing and able to maintain their usual diet (and, if indicated, maintain a lactose-free diet) during the course of the study.
6. All patients must have had either a full colonoscopy or flexible sigmoidoscopy with barium enema performed at some time in the past. Additionally, they must have these procedures repeated prior to the screening visit if:

   * the patient has experienced a recent change in bowel habits (recent means within 6 months of entry to the study) or
   * the patient is aged 55 or above (at their last birthday) and has not had these investigations carried out within 5 years of entry to the study.
7. Patients must be willing and able to comply with the study procedures.

Exclusion Criteria

A patient will be excluded from the study if any one of the following criteria applies to that patient:

1. Patients with severe concurrent disease defined as any disease which, in the investigator's opinion, is unstable and/or life-threatening, or is serious enough to jeopardize efficacy or safety assessments during the study. This definition may include, but is not limited to:

   * Any major GI disorder (including history of inflammatory bowel disease [colitis], celiac disease, complicated colonic diverticular disease)
   * History of abdominal surgery which, in the investigator's opinion, may interfere with the assessment of IBS symptoms during the study
   * Uncontrolled diabetes
   * Uncontrolled hypertension
   * Uncontrolled thyroid disease
   * History of cancer (with the exception of basal or squamous cell carcinoma)
   * A history of any serious psychiatric disorder (including schizophrenia, bipolar disorder [including current suicidal ideation or patients who have attempted suicide within 12 months of entry to the study] and any psychiatric disorder severe enough to warrant psychiatric hospital treatment, as an in-patient within 12 months of entry to the study)
2. Patients with current psychotic disorders, bipolar disorders, alcohol or drug dependence/abuse, anorexia nervosa or bulimia as identified by completing the Mini International Neuropsychiatric Interview at the screening visit.
3. Patients with clinically significant abnormal blood test results at entry to the study, in the opinion of the investigator.
4. Patients with anatomical lesions of the colon (except non-complicated diverticular disease) or microscopic colitis or inflammatory bowel disease as assessed by investigations carried out prior to the screening visit.
5. Patients with a history of lactose intolerance prior to the screening.
6. Patients with any history of drug or alcohol abuse in the past 6 months.
7. Patients on antidepressants for the treatment of mood or anxiety disorders.
8. Patients receiving any medication which may interfere with the assessment of IBS symptoms during the study, and which cannot be stopped. These medications include the following:

   * All antidepressant medication (including selective serotonin re-uptake inhibitors (SSRIs). Where antidepressant medication has been previously prescribed, the following timelines should be adhered to: a 42-day wash out period from Prozac™ (fluoxetine) before randomization into the study; a 2 week wash-out for other antidepressants.
   * Drugs with putative effect on transit (including, but not limited to, erythromycin, metoclopramide, cisapride, dicyclomine hydrochloride, hyoscyamine sulfate, etc.), anti-diarrheals (including, but not limited to dephenoloxilate with atropine, loperamide, bismuth, kaolin and pectin, etc.), and laxatives (oral or rectal). Bulking agents (including ispaghula husk, psyllium and dietary bran supplements) may be continued during the study, provided that the patient has been taking a stable dose for at lease 3 months prior to entering the study and that this dose does not change during the study. Patients taking bulking agents on an "as needed" basis must refrain from taking these medications during the study.
9. Patients who have taken an investigational drug within 30 days (or 5 half-lives, whichever is the longer) of entry to the study, or who are due to receive such a drug during the study.
10. Female patients who are pregnant or lactating.

The investigator should call the study monitor if he/she has any questions regarding patient eligibility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in: Changes in Mean composite pain scores (on IVRS) | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Associated symptoms of IBS (diarrhea, constipation, incomplete emptying, etc.) scores IBS Quality of Life scores Clinical Global Impression scores of 1 or 2 Beck Depression Inventory II Beck Anxiety Inventory | 12 weeks
Recording of spontaneous adverse events throughout the screening, run-in, and treatment phases of the study Conducting the DOTES at defined points during the study | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greg Clary, M.D., Principal Investigator — Duke University; Ashwin A Patkar, M.D., Principal Investigator — Duke University
Locations (1):
- Department of Psychiatry Clinical Trial Team, Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Marks DM, Han C, Krulewicz S, Pae CU, Peindl K, Patkar AA, Masand PS. History of depressive and anxiety disorders and paroxetine response in patients with irritable bowel syndrome: post hoc analysis from a placebo-controlled study. Prim Care Companion J Clin Psychiatry. 2008;10(5):368-75. doi: 10.4088/pcc.v10n0504. PMID 19158975